CLINICAL TRIAL: NCT05912842
Title: Forging Sustainable Solutions for HIV Continuity of Care Through Medical-legal Partnerships
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH125718 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Organizational Partnerships for Healthy Living; Standard of Care
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The investigative team will conduct a clustered-randomized small-scale trial in two HIV treatment services organizations in Philadelphia. One agency will be randomized to the OPAHL intervention, consisting of integrated legal support (n=100 PLWH) and one agency will be randomized to the standard of care, legal aid referral (n=100 PLWH).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Legal Partnerships (Experimental): Component 1 is a comprehensive training for all MLP care providers delivered to clinical, social and behavioral, and legal staff together to establish a collaborative environment. Component 2 consists of the screening tool and screening protocol that is designed to identify health-harming legal needs of PLWH patients. Component 3 includes the provision of legal support through partnership with the Legal Clinic for the Disabled. Upon a positive legal needs screening, the case manager connects the patient to this attorney, at which point the patient, after signing a letter of engagement, becomes a client and can now address the identified legal issue(s) with legal representation.
  Interventions: Behavioral: Organizational Partnerships for Healthy Living
- Standard of Care (Active Comparator): Comparison arm health organization will only receive the HIV standard of care (U.S. CDC HIV standard of care) and referral to legal aid.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Organizational Partnerships for Healthy Living — Component 1 is a comprehensive training for all MLP care providers delivered to clinical, social and behavioral, and legal staff together to establish a collaborative environment. Component 2 consists of the screening tool and screening protocol that is designed to identify health-harming legal needs of PLWH patients. Component 3 includes the provision of legal support through partnership with the Legal Clinic for the Disabled.
  Other Names: OPHAL
  Arms: Medical Legal Partnerships
Behavioral: Standard of Care — Comparison arm health organization will only receive the HIV standard of care (U.S. CDC HIV standard of care) and referral to legal aid.
  Arms: Standard of Care

SUMMARY:
The goal of this study is to test the Organizational Partnerships for Healthy Living (OPAHL) intervention through a feasibility and acceptability trial. OPAHL is an innovative, multilevel intervention package intended for health care organizations serving people living with HIV (PLWH). It was developed through a prior study (grant #: R21 MH115820) using intervention mapping methodology and community-scientific collaborative boards. OPAHL consists of: 1) training (7/8hours) for all MLP staff (clinical, social and behavioral services, and legal) on HIV continuum of care, health harming legal risks and needs, and MLP structure and operations to ensure that an integrated and collaborative environment is established from the earliest stages of the program; 2) case management training on the legal continuum of care; 3) embedding of legal expertise within regularized case management team meetings; 4) co-location of legal services in health care agencies through MLP inter-organizational partnership within 3 months; and 5) organizationally tailored implementation of best-practice communication and information-sharing protocols among providers within MLP, anchored in patient autonomy and choice. The specific aims of this study are: 1) to refine the OPAHL intervention prototype for implementation with PLWH with detectable viral loads and 2) to test the feasibility, acceptability and preliminary effects sizes of OPAHL. Given the current COVID-19 pandemic, the study will also explore MLP opportunities that respond at the intersection of HIV/AIDS and COVID-19 prevention and treatment.

DETAILED DESCRIPTION:
A health-harming legal need is a social problem that adversely affects a person's health or access to health care and which is better remedied through the combination of legal care and health care. Medical legal partnerships (MLPs) have been underutilized as structural interventions; however, they could help improve HIV care continuum outcomes in health care organizations. The goal of this study is to test the Organizational Partnerships for Healthy Living (OPAHL) intervention through a feasibility and acceptability trial. OPAHL is an innovative, multilevel intervention package intended for health care organizations serving people living with HIV (PLWH). It was developed through a prior study (grant #: R21 MH115820) using intervention mapping methodology and community-scientific collaborative boards. OPAHL consists of: 1) training (7/8hours) for all MLP staff (clinical, social and behavioral services, and legal) on HIV continuum of care, health harming legal risks and needs, and MLP structure and operations to ensure that an integrated and collaborative environment is established from the earliest stages of the program; 2) case management training on the legal continuum of care; 3) embedding of legal expertise within regularized case management team meetings; 4) co-location of legal services in health care agencies through MLP inter-organizational partnership within 3 months; and 5) organizationally tailored implementation of best-practice communication and information-sharing protocols among providers within MLP, anchored in patient autonomy and choice. The specific aims of this study are: 1) to refine the OPAHL intervention prototype for implementation with PLWH with detectable viral loads and 2) to test the feasibility, acceptability and preliminary effects sizes of OPAHL. Given the current COVID-19 pandemic, the study will also explore MLP opportunities that respond at the intersection of HIV/AIDS and COVID-19 prevention and treatment. Two health care organizations serving PLWH Philadelphia, PA that do not currently provide any form of legal services to their patients will participate in this trial (n=200 PLWH). The proposed study is in response to PA-20-141: Formative and Pilot Intervention Research for Prevention and Treatment of HIV/AIDS (R34 Clinical Trial Optional). It is also responsive to two of the areas of high priority research of NIMH Division of AIDS Research (Develop and test interventions to improve HIV treatment outcomes; Advance the development and testing of interventions delivered beyond the individual level). Completion of this project will result in the development of an intervention package to optimize HIV services for a highly vulnerable population whose HIV care is affected by health-harming legal needs.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV (as confirmed by medical record)
* 18 years or older
* HIV viral load of more than 200 copies/mL (as confirmed by medical record)
* Willing and able to consent to participate in the trial (including accessing their medical records at the health care organization)
* No intent to relocate within the 6 months following their enrollment in the study

Exclusion Criteria:

-Individuals who self-report having been sentenced to serve under state or federal custody, with a sentence to begin within 6 months from proposed enrollment in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression | 6 months
  HIV viral load through HIV Nucleic Acid Amplification Test (NAAT) HIV by PCR HIV RNA Test

SECONDARY OUTCOMES:
Engagement in HIV Care | 6 months
  HIV primary care appointments and services at health organization (Attendance in the prior 3 months)
Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 | 6 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 is a gauge of general healthcare-related quality of life.Response options are presented as 5-point (as well as a single 11-point) rating scales. The scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.

CONTACTS AND LOCATIONS:
Locations (1):
- TPAC, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided